CLINICAL TRIAL: NCT06638619
Title: Comparative Efficacy of Saccadic and Biofeedback Training in Homonymous Hemianopia: A Comprehensive Eye Movement Pilot Study
Brief Title: Comparative Efficacy of Saccadic and Biofeedback Training in Homonymous Hemianopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jason Eugene Vice, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013228; 000 (Other Grant/Funding Number: Vision Science Research Center)
Record Dates: First submitted 2024-09-30; First posted 2024-10-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hemianopia, Homonymous
Keywords: stroke; vision; hemianopia
MeSH Terms: conditions — Hemianopsia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback Fixation Arm (Experimental): Biofeedback training is a mind-body therapy that helps people learn to control their involuntary bodily functions, such as eye movements. The goal is to improve eye movement control to improve gaze stability.
  Interventions: Behavioral: Biofeedback Fixation Training
- Saccadic Reading Arm (Active Comparator): Saccadic reading training helps people to learn to control their involuntary eye movements. The goal is to improve eye movement control to improve saccadic and fixational behaviors during reading activities.
  Interventions: Behavioral: Saccadic Reading Training

INTERVENTIONS:
Behavioral: Biofeedback Fixation Training — This training type involves the use of microperimetry. Microperimetry is a visual field test that incorporates perimetry and retinal imaging and is a standard ophthalmic clinical technology. It allows for direct observation of the fundus, but uses an eye-tracking system to compensate for involuntary eye movements. A program designed to train patients to direct and hold their gaze at an eccentric location programmed by the controller will be used. When the participant directs their gaze towards the pre-programmed location, a sound of increasing frequency is emitted to let them know they are approaching the correct location. The sound stabilizes into a solid tone when the patient is gazing directly at the trained location (biofeedback) and they are asked to attempt to hold their gaze at this location for as long as possible.
  Arms: Biofeedback Fixation Arm
Behavioral: Saccadic Reading Training — Participants will be assigned to participate in an at-home reading program. The reading exercises consist of worksheets with letter and number combinations of increasing complexity and font sizes. They are intended to increase accuracy in identifying letters and numbers. Worksheets will initially be dispensed with larger font type and spacing and be graded at weekly intervals towards regular, newspaper-size print and spacing over the course of training.
  Arms: Saccadic Reading Arm

SUMMARY:
This pilot study aims to understand how eye movements change in people with vision loss from stroke after completing one of two types of training. The study will look at how eye movements and reading performance change after training. Researchers will compare the results of two groups: one group will complete five clinical training sessions using an eye-tracking machine for 30 minutes each, while the other group will do at-home reading exercises for 20 minutes a day, 5 days a week, for 6 weeks. The goal is to see if there is a difference in performance between the two types of training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* Presence of hemianopia with central vision involvement
* Stroke occurred at least 6-months before enrollment

Exclusion Criteria:

* Presence of hemianopia with macular sparing
* Diagnosis of hemispatial neglect

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Oculomotor Metrics | Pre-training and at 6-weeks.
  Participants will be asked to read aloud a series of sentences presented on a display. Eye movements will be recorded in real-time using an Eye-Link 1000 infrared eye-tracking camera, as the patient is reading what is on the display. The primary outcome measure will be the first saccade landing location.

SECONDARY OUTCOMES:
Pepper Visual Skills Reading Test (VSRST) | Pre-training and at 6-weeks.
  A clinical reading assessment used in low vision settings to assess for common patterns of reading errors (misidentifications, skipped letters or words, skipped lines). The participant reads aloud lines of text (random letters and words of increasing complexity and decreasing line spacing.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Vice, Ph.D., Principal Investigator — University of Alabama at Birmingham